CLINICAL TRIAL: NCT01817452
Title: A Prospective, Randomized Multicenter, Open-label Comparison of Preoperative Combination of Trastuzumab and Pertuzumab With or Without Concurrent Taxane Chemotherapy Given for Twelve Weeks in Patients With Operable HER2+/HR- Breast Cancer Within the ADAPT Protocol
Acronym: ADAPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM06 / ADAPT HER2+/HR-
Record Dates: First submitted 2013-03-18; First posted 2013-03-25 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Trastuzumab + Pertuzumab
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab
- Arm B (Active Comparator): Trastuzumab + Pertuzumab + Paclitaxel
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Trastuzumab
  Other Names: Herceptin
Drug: Pertuzumab
Drug: Paclitaxel
  Arms: Arm B

SUMMARY:
Trial to evaluate efficacy of dual blockade with two anti-HER2 agents with or without chemotherapy backbone within the ADAPT trial.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age at diagnosis 18 years and above (consider patients at 70 years and above for ADAPT Elderly)
* Histologically confirmed unilateral primary invasive carcinoma of the breast
* Clinical T1 - T4 (except inflammatory breast cancer)
* All clinical N (cN)
* No clinical evidence for distant metastasis (M0)
* Known HR status and HER2 status (local pathology) Tumor block available for central pathology review
* Performance Status ECOG ≤ 1 or KI ≥ 80%
* Negative pregnancy test (urine or serum) within 7 days prior to start of induction treatment in premenopausal patients
* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
* The patient must be accessible for treatment and follow-up

Additional Inclusion criteria for participation in the HR-/HER2+ sub-protocol:

* Confirmed ER and PR negative and HER2+ by central pathology
* Clinical cT1c - T4a-c (participation of patients with tumors >cT2 is strongly recommended)
* All clinical N (participation of patients with cN0, if at least cT1c is strongly recommended)
* Patients must qualify for neoadjuvant treatment
* LVEF > 50%; LVEF within normal limits of each institution measured by echocardiography and normal ECG (within 42 days prior to induction treatment)

Exclusion Criteria:

* Known hypersensitivity reaction to the compounds or incorporated substances
* Prior malignancy with a disease-free survival of < 10 years, except curatively treated basalioma of the skin, pTis of the cervix uteri
* Non-operable breast cancer including inflammatory breast cancer
* Previous or concurrent treatment with cytotoxic agents for any reason after consultation with the sponsor
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry
* Male breast cancer
* Concurrent pregnancy; patients of childbearing potential must implement a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
* Breast feeding woman
* Sequential breast cancer
* Reasons indicating risk of poor compliance Patient not able to consent

Additional Exclusion Criteria for participation in the HER2+/HR- sub-protocol:

* Known polyneuropathy ≥ grade 2
* Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study
* Inadequate organ function (e.g. hepatic impairment, pulmonary disease, etc.)
* Uncompensated cardiac function (current unstable ventricular arrhythmia requiring treatment, history of symptomatic CHF NYHA classes II-IV), history of myocardial infarction or unstable angina pectoris within 6 months of enrollment, history of severe hypertension, CAD - coronary artery disease)
* Severe dyspnea
* Abnormal blood values:
* Thrombocytopenia > CTCAE grade 1
* Increases in ALT/AST > CTCAE grade 1
* Hypokalaemia > CTCAE grade 1
* Neutropenia > CTCAE grade 1
* Anaemia > CTCAE grade 1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Definition of a biomarker (profile) characterizing "good responders" to dual blockade T and P anti-HER2 blockade that have similar pCR rates as patients treated with identical dual anti-HER2 blockade + taxane backbone | After 12 weeks of therapy
  pCR will be measured after 12 weeks of randomized treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr., Principal Investigator — Breast Center of the University of Munich (LMU), Universitätsfrauenklinik Großhadern, Munich, Germany; Ulrike Nitz, Prof. Dr., Study Chair — Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, Germany
Locations (1):
- Ev. Krankenhaus Bethesda Brustzentrum Niederrhien, Mönchengladbach, Germany

REFERENCES:
- [Background] Hofmann D, Nitz U, Gluz O, Kates RE, Schinkoethe T, Staib P, Harbeck N. WSG ADAPT - adjuvant dynamic marker-adjusted personalized therapy trial optimizing risk assessment and therapy response prediction in early breast cancer: study protocol for a prospective, multi-center, controlled, non-blinded, randomized, investigator initiated phase II/III trial. Trials. 2013 Aug 19;14:261. doi: 10.1186/1745-6215-14-261. PMID 23958221
- [Derived] Graeser M, Gluz O, Biehl C, Ulbrich-Gebauer D, Christgen M, Palatty J, Kuemmel S, Grischke EM, Augustin D, Braun M, Potenberg J, Wuerstlein R, Krauss K, Schumacher C, Forstbauer H, Reimer T, Stefek A, Fischer HH, Pelz E, Zu Eulenburg C, Kates R, Ni H, Kolberg-Liedtke C, Feuerhake F, Kreipe HH, Nitz U, Harbeck N. Impact of RNA Signatures on pCR and Survival after 12-Week Neoadjuvant Pertuzumab plus Trastuzumab with or without Paclitaxel in the WSG-ADAPT HER2+/HR- Trial. Clin Cancer Res. 2023 Feb 16;29(4):805-814. doi: 10.1158/1078-0432.CCR-22-1587. PMID 36441798
- [Derived] Nitz U, Gluz O, Graeser M, Christgen M, Kuemmel S, Grischke EM, Braun M, Augustin D, Potenberg J, Krauss K, Schumacher C, Forstbauer H, Reimer T, Stefek A, Fischer HH, Pelz E, Zu Eulenburg C, Kates R, Wuerstlein R, Kreipe HH, Harbeck N; WSG-ADAPT investigators. De-escalated neoadjuvant pertuzumab plus trastuzumab therapy with or without weekly paclitaxel in HER2-positive, hormone receptor-negative, early breast cancer (WSG-ADAPT-HER2+/HR-): survival outcomes from a multicentre, open-label, randomised, phase 2 trial. Lancet Oncol. 2022 May;23(5):625-635. doi: 10.1016/S1470-2045(22)00159-0. Epub 2022 Apr 8. PMID 35405088
- [Derived] Graeser M, Schrading S, Gluz O, Strobel K, Herzog C, Umutlu L, Frydrychowicz A, Rjosk-Dendorfer D, Wurstlein R, Culemann R, Eulenburg C, Adams J, Nitzsche H, Prange A, Kummel S, Grischke EM, Forstbauer H, Braun M, Potenberg J, von Schumann R, Aktas B, Kolberg-Liedtke C, Harbeck N, Kuhl CK, Nitz U. Magnetic resonance imaging and ultrasound for prediction of residual tumor size in early breast cancer within the ADAPT subtrials. Breast Cancer Res. 2021 Mar 18;23(1):36. doi: 10.1186/s13058-021-01413-y. PMID 33736679